CLINICAL TRIAL: NCT02826707
Title: Feasibility Evaluation of a Smartphone-delivered Peer-led Physical Activity Counselling Program for Improving Physical Activity in Manual Wheelchair Users
Brief Title: Evaluation of a Smartphone-delivered Peer-led Physical Activity Counselling Program for Manual Wheelchair Users
Acronym: ALLWheel
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: McGill University (Other)
Responsible Party: Principal Investigator, Krista Best, Assistant Professor/ Researcher, Laval University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SPPAC2016
Record Dates: First submitted 2016-05-31; First posted 2016-07-11 (Estimated); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Physical Activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SPPAC intervention (Experimental): Smartphone-delivered peer-led physical activity counselling
  Interventions: Behavioral: SPPAC intervention
- Control group (No Intervention): Pragmatic no-contact control group

INTERVENTIONS:
Behavioral: SPPAC intervention — A peer coach will deliver a physical activity counselling intervention using a Smartphone. Individualized programs will be based on participants physical activity/wheelchair mobility goals.
  Arms: SPPAC intervention

SUMMARY:
Despite physical activity (PA) being a valuable modality for promoting health, the evidence for effective PA intervention strategies for manual wheelchair (MWC) users is underdeveloped. Community-based programs and telephone-counselling interventions to increase PA among MWC users have had some success, but the uptake and adherence to these interventions remains low within this population. Community-based programs may not reach MWC users who live in rural areas and have issues with transportation, while health professionals may not optimally relate with MWC when providing telephone counselling. Although the PA needs of MWCs are not fully understood, there is reason to believe that including peers into intervention delivery may have benefits.

A feasibility trial is critical and prudent prior to moving forwards with a large and expensive multi-site randomized controlled trial (RCT) to ensure that: the intervention meets the needs of the target population; the right outcomes are measured; and that the intervention is feasible to administer.

The objective of this study is to evaluate the feasibility of a Smartphone-delivered Peer-led Physical Activity Counselling (SPPAC) program for MWC users.

ELIGIBILITY:
Inclusion Criteria:

* live in the community
* have used a manual wheelchair for ≥ 1 year
* able to self-propel a manual wheelchair for at least 10m
* able to communicate in English or French
* have physical activity or mobility goals
* cognitively able to set goals (Mini-mental State Exam Score ≥ 25)

Exclusion Criteria:

* anticipate a health condition or procedure that contraindicates training (e.g., surgery scheduled which would impair physical activity)
* have a degenerative condition that is expected to progress quickly (e.g., Amyotrophic Lateral Sclerosis
* are concurrently or planning to receive manual wheelchair mobility training over the period of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-02-07 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Objective physical activity | Change in physical activity from baseline to post-intervention (10 weeks post-baseline) and at follow-up (3 months post-intervention
  Physical activity will be measured objectively using Actigraphy, a small, lightweight accelerometry-based tri-axial activity monitor (Actigraph 3GTX) that is worn on the wrist and MWC without impeding bodily movements or PA. Information about motion direction and speed are integrated to produce an electrical current with variable magnitude and duration. The electrical current data are stored in the monitor as 'activity counts.'

SECONDARY OUTCOMES:
Subjective physical activity (Leisure-Time Physical Activity Questionnaire (LTPA)) | Change in LTPA from baseline to post-intervention (10 weeks post-baseline) and at follow-up (3 months post-intervention
  Self-reported frequency (number of bouts) and duration (min per bout) of light, moderate and heavy intensity PA over the past 7 days.
Wheelchair skills capacity and performance (Wheelchair Skills Test- Questionnaire (WST-Q)) | Change in WST from baseline to post-intervention (10 weeks post-baseline) and at follow-up (3 months post-intervention
  Subjective evaluation of the skills capacity and performance of 32 manual wheelchair skills.
Physical activity motivation (Behavioural Regulation in Exercise Questionnaire (BREQ-2)) | Change in BREQ-2 from baseline to post-intervention (10 weeks post-baseline) and at follow-up (3 months post-intervention
  Subjective evaluation of motivation for physical activity is measured using 5 subscales of regulation: external, introjected identified, intrinsic and amotivation.
Perceived autonomy support (Health Care Climate Questionnaire (HCCQ)) | Change in HCCQ from baseline to post-intervention (10 weeks post-baseline) and at follow-up (3 months post-intervention
  Subjective evaluation of perceived autonomy support
Satisfaction of psychological needs (Psychological Need Satisfaction in Exercise Scale (PNSES)) | Change in PNSES from baseline to post-intervention (10 weeks post-baseline) and at follow-up (3 months post-intervention
  Subjective evaluation of satisfaction of psychological needs (i.e. autonomy, competence, relatedness) for physical activity will be measured only in the intervention group.
Self-efficacy to overcome barriers to leisure-time physical activity (Leisure-time Physical Activity Barrier Self-efficacy Scale) | Change in Self-efficacy to overcome barriers to leisure-time physical activity from baseline to post-intervention (10 weeks post-baseline) and at follow-up (3 months post-intervention
  Subjective evaluation of self-efficacy to overcome salient barriers to physical activity participation (e.g. when faced with transportation problems, bad weather, pain and fatigue).
Wheelchair use self-efficacy (Wheelchair Use Confidence Scale Short Form (WheelCon-SF)) | Change in WheelCon-SF from baseline to post-intervention (10 weeks post-baseline) and at follow-up (3 months post-intervention
  Subjective evaluation of situations that challenge self-efficacy while using a manual wheelchair.
Satisfaction with participation in physical activity using a wheelchair (Wheelchair Outcome Measure (WhOM)) | Change in WhOM from baseline to post-intervention (10 weeks post-baseline) and at follow-up (3 months post-intervention
  A semi-structured interview that allows participants to select important physical activity/wheelchair mobility participation goals. The importance and current level of satisfaction is evaluated.
Measure of self-efficacy in performing functional activities of daily living in individuals with Spinal Cord Injury (Moorong Self Efficacy Scale - MSES) | Change in MSES from baseline to post-intervention (10 weeks post-baseline) and at follow-up (3 months post-intervention
  Subjective evaluation of self-efficacy in carrying out activities of daily living. Minimum value 1 and maximum value 7. A higher score indicates a higher perceived self efficacy.
Measure the degree to which individuals who have experienced traumatic or incapacitating illness achieve reintegration into normal social activities (Reintegration to Normal Living Index - RNLI) | Change in RNLI from baseline to post-intervention (10 weeks post-baseline) and at follow-up (3 months post-intervention
  Subjective evaluation of the reintegration to normal living activities

CONTACTS AND LOCATIONS:
Overall Officials: François Routhier, PhD, Principal Investigator — Laval University
Locations (1):
- Centre for Interdisciplinary Research in Rehabilitation and Social Integration, Québec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Best KL, Routhier F, Sweet SN, Arbour-Nicitopoulos KP, Borisoff JF, Noreau L, Martin Ginis KA. The Smartphone Peer Physical Activity Counseling (SPPAC) Program for Manual Wheelchair Users: Protocol of a Pilot Randomized Controlled Trial. JMIR Res Protoc. 2017 Apr 26;6(4):e69. doi: 10.2196/resprot.7280. PMID 28446419